CLINICAL TRIAL: NCT06544941
Title: Improving Maternal Mental Health in Military-Affiliated Pregnant Women: Effectiveness of a Smart Bassinet
Brief Title: Improving Maternal Sleep and Mental Health
Acronym: SHINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Collaborators: University of Virginia (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HT94252410690
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-08

CONDITIONS: Postpartum Depression; Postpartum Anxiety; Sleep Disturbance; Infant Behavior; Maternal Behavior; Inflammation; Military Family
Keywords: sleep; postpartum; intervention; inflammation; depression; anxiety
MeSH Terms: conditions — Depression, Postpartum; Parasomnias; Infant Behavior; Inflammation; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Women are randomized to one of two bassinets to use for up to 6 months PP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Smart Bassinet (SB) (Experimental): The SB responds to an infant who is fussing or crying by initiating "swaying" movement and "shushing" sounds with white noise that incrementally increase until the infant calms or the caregiver shuts it off. It will help babies transition into life outside of the womb with ease, enabling them to feel safe and secure, which translates to more sleep.
  Interventions: Device: Smart Bassinet
- HALO Bassinet (TAU) (Active Comparator): The HALO is a commercially available bassinet that does not have any robotic/responsive actions incorporated within it.
  Interventions: Device: HALO

INTERVENTIONS:
Device: Smart Bassinet — The SNOO will respond to a crying or fussing infant in order to soothe and calm it down.
  Other Names: Robotic, responsive bassinet, SNOO
  Arms: Smart Bassinet (SB)
Device: HALO — The HALO is a commercially available bassinet
  Arms: HALO Bassinet (TAU)

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a Smart Bassinet to prevent/mitigate postpartum mood disorders by augmenting maternal sleep and/or enhancing infant sleep. The investigators will conduct a 2-arm randomized controlled trial (RCT) to compare infant and maternal sleep of infants who use a smart bassinet (SB) or a standard commercially available bassinet (Halo Bassinest Swivel Sleeper 3.0) (usual/traditional care (TAU)). After confirmation of eligibility, participants (N = 342) will randomly be assigned to either the SB or TAU. The investigators hypothesize that use of the SB will be associated with better infant and maternal sleep over a 6-month period, and these mothers will report fewer depressive and anxiety symptoms across the postpartum. The main question[s] it aims to answer [is/are]:

Aim 1: Determine the effect of the SB on infant sleep and maternal sleep. [primary hypothesis or outcome measure 2]? Aim 2: Determine the effect of the SB on maternal postpartum depressive symptoms and evaluate the model that the association between the SB and postpartum depressive symptoms is mediated by both infant and maternal sleep Aim 3: Compare trajectory of immune system function from late pregnancy through postpartum between PPD and non-PPD and between SB and TAU groups Exploratory Aim. Evaluate whether the elevated risk demonstrated by previously identified PPD epigenetic biomarkers at the TTC9B and HP1BP3 genes can be modified by using a SB. The investigators hypothesize that the elevated risk will be reduced in the SB condition compared to TAU.

Military-affiliated pregnant women will be recruited from across the US via social media and advertising. Monthly online questionnaires will be completed by the mother. Objective sleep data will be collected monthly using an actigraph for 1-week from both mother and baby. Blood samples for assay of inflammatory markers will be collected at enrollment, 3- and 6- months postpartum.

DETAILED DESCRIPTION:
The investigators propose to conduct a 2-arm randomized controlled trial (RCT) to compare infant and maternal sleep of infants who use the SB or a standard commercially available bassinet (Halo Bassinest Swivel Sleeper 3.0) (usual/traditional care (TAU)).

The primary objective of this proposal is to randomly assign mother-infant dyads (N = 342) to the SB or the TAU condition and follow them monthly for 6 months. Mothers will complete online surveys monthly regarding infant sleep and behavior, maternal sleep, and maternal depressive symptoms. Prospective subjective and objective sleep data will also be collected from mother and infant for one week each month. This study represents the first empirical study to assess the efficacy of the SB to promote efficient infant sleep, and to assess longitudinal effects on maternal postpartum sleep and mood symptoms. This work is essential since few effective interventions are available that support infant sleep. A secondary objective is to explore maternal biomarkers of PPD, including markers of inflammation and epigenetic biomarkers, and determine if the SB intervention alters immune dysregulation and the risk associated with epigenetic biomarkers of PPD. The rationale stems from evidence regarding dysregulation of the immune system and inflammatory activity as potential mediating pathways between sleep disturbances and health.

This proposal will address the following aims:

Aim 1: Determine the effect of the SB on infant sleep and maternal sleep. Hypothesis 1a: Infants who sleep in the SB will have better sleep (i.e., diary and Brief Infant Sleep Questionnaire as maternally reported) compared to TAU. Outcomes will include maternally reported sleep duration, awakenings, as well as objective assessed (actigraphy) wake after sleep onset (WASO), and sleep onset latency (SOL). Hypothesis 1b: Mothers of infants who sleep in the SB will have better subjectively reported (i.e., diary and Pittsburgh Sleep Quality Index) and objectively assessed (actigraphy) sleep compared to TAU. Outcomes will be the same as the infants.

Aim 2: Determine the effect of the SB on maternal postpartum depressive symptoms and evaluate the model that the association between the SB and postpartum depressive symptoms is mediated by both infant and maternal sleep. Hypothesis 2a: Mothers of infants who sleep in the SB will have fewer postpartum depressive symptoms over time (i.e., Edinburgh Postnatal Depression Scale) compared to TAU. Hypothesis 2b: The SB improves infant sleep, which then predicts better maternal sleep, and thereby predicts lower maternal depressive symptoms.

Aim 3: Compare trajectory of immune system function from late pregnancy through postpartum between PPD and non-PPD and between SB and TAU groups. Hypothesis 3: Peripheral cytokines, immune cells, and stimulated cytokine profiles of women with PPD assessed in late pregnancy, 3- and 6- months postpartum, will indicate greater innate immune activity compared to those who do not develop PPD. Hypothesis 3b: Mothers of infants who sleep in the SB will exhibit less innate immune dysfunction than TAU mothers.

Exploratory Aim. Evaluate whether the elevated risk demonstrated by previously identified PPD epigenetic biomarkers at the TTC9B and HP1BP3 genes can be modified by using a SB. The investigators hypothesize that the elevated risk will be reduced in the SB condition compared to TAU.

Participants. Eligible Pregnant women (N = 342) will be enrolled and randomly assigned to SB or TAU stratified by epigenetic status in the late 3rd trimester and followed longitudinally every month for 6 months. Inclusion criteria: History of depression; singleton gestation; 18-45 years of age; ability to communicate during the screening process; access to a computer, responsive phone, or tablet with internet service; and willing to use the bassinet they are randomized to. Exclusion criteria: clinical confirmation of any current psychopathology (depression, anxiety, suicidal intent, bipolar disorder, etc.), use of psychotropic or sleep medications, multiple gestations, pregnancy/birth complications that would interfere with bassinet use, plans to co-sleep with infant exclusively, tobacco, alcohol, or substance abuse during pregnancy. Self-reported, untreated comorbid sleep disorders, including narcolepsy, periodic leg movement disorder, and/or obstructive sleep apnea.

Initial clinical assessment of depression: Psychopathology will be assessed over the phone using The Structured Clinical Interview for DSM-5 Disorders (SCID-5-CV).

Randomization. Mothers-infant dyads (up to N = 342) will be randomly assigned to conditions by using a random number generating program found on a widely used and reputable website (www.randomizer.org)". This will further allow for comparability between the SB and current usual care/common sleep arrangements. The investigators will perform 1:1 randomization, stratifying for epigenetic status. The SB will be shipped to participants and returned at the expense of Happiest Baby, Inc. TAU participants will be shipped the Halo Bassinest Swivel Sleeper bassinet.

Data Collection. For each assessment, all participants will receive an email with a REDCap link for online data collection. To mitigate and minimize the possibility of missing data in the measures, electronic questionnaires will be programmed to prevent skipping questions. In addition, participants will receive a monthly package containing two actigraphs, maternal sleep diaries, the Baby's Day Diary, a certified blood mailer with tubes, and a prepaid return envelope.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a singleton gestation who have a military affiliation
* Ages 18-45 years
* Ability to communicate during the screening process
* Access to a computer, smart phone or tablet with internet service
* Willing to use bassinet they are randomized to
* Willing to travel to a local Quest for blood draw

Exclusion Criteria:

* Presence of depression assessed over the phone using the Structured Clinical Interview for DSM Disorders - Clinical Version, Mood Disorders Section (SCID-I). Current active suicidal ideation, medical or psychiatric instability, or active substance abuse or dependence during the last 90 days. Since this is a study about risk for recurrent PPMD, actively depressed women will be excluded.
* Plans to co-sleep with infant. The goal is to compare two bassinets; therefore co-sleeping would prohibit extensive use of a bassinet.
* Under the age of 18 years or > 45 years. The goal is to include women of childbearing age.
* Multiple gestations, Type 1 diabetes, congenital fetal anomalies. Women with these factors will likely have major disruption of sleep, require 2 bassinets, or a disrupted home life. These would skew the data and make interpretations and comparisons difficult.
* Tobacco use (current). Smoking is associated with poor sleep and inflammation.
* Self-reported, untreated comorbid sleep disorders including narcolepsy, periodic leg movement disorder, and/or obstructive sleep apnea. These disorders contribute to poor sleep and often require medications for treatment.
* Current use of psychotropic or sleep medications. These are associated with altered sleep and inflammation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 342 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Maternal Mood | 0-6 months postpartum
  Assessment of depressive and anxiety symptoms across the first 6 months postpartum
Maternal Sleep | 0-6 months postpartum
  Assessment of sleep across the first 6 months postpartum
Infant Sleep | 0-6 months postpartum
  Assessment of infant sleep across the first 6 months postpartum
Maternal Inflammation | late pregnancy, 3 & 6 months postpartum
  Assessment of changes in maternal inflammation

SECONDARY OUTCOMES:
Epigenetic biomarkers at the TTC9B and HP1BP3 genes | assess markers at Baseline (Late pregnancy)
  Evaluate whether the elevated risk previously demonstrated can be modified by using a SB.

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Okun, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- University of Colorado Colorado Springs, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The degree to which we share will be based on the US Army's decision.

REFERENCES:
- [Derived] Okun ML, Payne JL, Osborne LM, Feliciano L, Lac A. Effects of Using a Smart Bassinet on the Mental Health of Military-Affiliated Pregnant Women: Protocol for a Randomized Controlled Sleep Health and Mood in Newly Expectant Military Mothers (SHINE) Trial. JMIR Res Protoc. 2025 Apr 10;14:e66439. doi: 10.2196/66439. PMID 40209215